CLINICAL TRIAL: NCT04633590
Title: Effects of Home-based Exercise Gaming on Cardio-Metabolic and Cognitive Health Markers in Physically Inactive Individuals
Brief Title: Home-Based Exercise Gaming for Physically Inactive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HomeExergame
Record Dates: First submitted 2020-11-10; First posted 2020-11-18 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Physical Inactivity
Keywords: Home-based exercise gaming; Cardiovascular health; Neurocognitive health; Physical Inactivity; Exergame
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A single-centre, single-armed, open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- home-based exergaming (Experimental): The home-based exergame intervention will take place in an unsupervised place of the participant's choosing. Participants will be provided with all of the equipment (including a television if required) and receive instructions on how to use the system. Participants will be provided with a stepped training plan with exergame session durations of 19 minutes (4x 3-minutes 45-seconds of exercise interspersed with 1 minute of rest) in weeks 1 and 2; 24-minutes (4x 5-minutes of exercise interspersed with 1 minute of rest) in week 3 and 4; and 30-minutes (5x 5-minutes of exercise interspersed with 1 minute of rest) in week 5 and 6. Sessions will be set at a vigorous intensity (≥80% heart rate maximum) and participants will be provided with individualised heart rate zones to achieve in line with heart rate maximum determined during a maximal exercise test in Visit 2. Participants will be asked to train 3 times per week.
  Interventions: Behavioral: Home-based exergaming

INTERVENTIONS:
Behavioral: Home-based exergaming — Participants will undertake one of two 6-week training interventions. In both groups participants will be asked to train 3 times per week (18 sessions total), during which adherence to the training will be measured. To monitor adherence to training and training load (exercise completion, exercise duration and heart rate achieved during workouts) throughout the 6 weeks participants will be given a heart rate monitor.

SUMMARY:
Current guidelines recommend that adults undertake at least 150 minutes of moderate intensity physical activity or 75 minutes of vigorous physical activity per week. However, many adults fail to be physically active according to this definition of the World Health Organisation (WHO). This represents a large economic burden to healthcare systems and public health. A number of behavioural and environmental factors associated with modern lifestyles are largely responsible for the high levels of physical inactivity including; motorised transport and sedentary jobs, lack of time, limited access to adequate exercise facilities, lack of motivation, financial constraints and environmental factors including bad weather. In an attempt to overcome many of the common barriers to exercise, members of our research group developed a virtually-monitored exercise intervention that used simple on-the-spot bodyweight exercises to be performed in the participant's home without supervision or equipment. This home-based intervention was designed to be a practical and effective training strategy capable of producing metabolic and functional adaptions while removing many of the common barriers to exercise. Despite promising results, more engaging exercise strategies are needed to motivate sedentary individuals to increase their physical activity.

Inspired by current trends in the fitness market, Sphery Ltd. developed an immersive and motivating fitness exercise game (exergame), the "ExerCube". The ExerCube allows a full-body workout that concurrently challenges physical and cognitive functions and adapts to the fitness and skill level of the individual. The development of a home-based version of the ExerCube has the potential to make this system available to more individuals, reduce major barriers to exercise, and ultimately provide a strategy to improve cardio-metabolic health in the population. Innovative home-based exergames are particularly in demand given the increase in the number of people wanting to exercise at home due to the COVID-19 pandemic.

DETAILED DESCRIPTION:
Current guidelines recommend that adults undertake at least 150 minutes of moderate intensity physical activity or 75 minutes of vigorous physical activity per week. Regular physical activity improves many cardiovascular and metabolic health makers including beneficial effects on body weight, insulin sensitivity, glycaemic control, lipid profile, endothelial function and aerobic capacity. Despite overwhelming evidence that an inactive lifestyle leads to chronic disease and premature death, many adults fail to meet physical activity guidelines. Physical inactivity, defined as physical activity levels less than those required for optimal health and prevention of premature death, is a public health crisis. More than 1.4 billion adults worldwide classed as physically inactive, representing a large economic burden to healthcare systems. Clearly, new strategies are urgently needed to increase physical activity participation in the increasingly inactive population.

A number of behavioural and environmental factors associated with modern lifestyle including urbanisation, mechanisation and increased motorised transport are largely responsible for the high prevalence of physical inactivity, in addition to a number of common exercise barriers. Lack of time is cited as the main barrier to exercise as many individuals feel that increasing work hours and family commitments mean they cannot achieve the physical activity guidelines. Other common barriers within the general population include limited access to exercise facilities and appropriate equipment, difficulty with transportation, inadequate financial resources, bad weather and lack of motivation to engage in regular exercise. In an attempt to overcome many of the common barriers to exercise, members of our research group developed a virtually-monitored exercise intervention that used simple on-the-spot bodyweight exercises that could be performed in the participant's home without supervision or equipment. This home-based intervention was designed to be a practical and effective training strategy capable of producing metabolic and functional adaptions while removing many of the common barriers to exercise uptake and adherence such as "intimidating" gym environments, difficulty with access to facilities, travel time and financial constraints. Although these pilot studies successfully reduced common exercise barriers, more engaging exercise strategies are needed to increase levels of physical activity in the physically inactive population.

Inspired by current trends in the fitness market, the Swiss company Sphery Ltd. developed an immersive and motivating fitness exercise game (exergame), the "ExerCube". The ExerCube provides a full-body workout that concurrently challenges physical and cognitive functions as well as adapting to the individuals' fitness and skill level. Previous research has shown that the ExerCube is an effective training method that is more enjoyable than conventional exercise training. Development of a home-based version of the ExerCube has the potential to make this system available to more individuals, and to reduce major barriers to exercise, providing an attractive strategy to improve cardio-metabolic health of the population. Innovative home-based exergames are in demand given the increase in the number of people wanting to exercise at home due to the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-55
* Physically inactive, defined as not meeting the exercise guidelines of 150 minutes of moderate physical activity or 75 minutes of vigorous physical activity per week
* BMI 18.5 kg/m2 - 30 kg/m2
* No known cardiovascular disorders
* Able to provide written informed consent and understand instructions

Exclusion Criteria:

* Overt diabetes mellitus (type 1, type 2, other forms of diabetes)
* Pregnant, planning on becoming pregnant during the study, or breast feeding
* Physical or psychological disease likely to interfere with the normal conduct of the study as judged by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
VO2max | Pre to post 6 weeks of home-based exergame training
  Change in maximal aerobic capacity (VO2max)

SECONDARY OUTCOMES:
Wmax | Pre to post 6 weeks of home-based exergame training
  Change in maximal power output (Wmax)
Adherence | 6 weeks of home-based exergame training
  Training adherence indicated by the number of training sessions performed over the 6 week period
Adherence | 6 weeks of training
  Training adherence indicated by the number of training sessions in which the desired exercise intensity was achieved over the 6 week period
Drop-out rate | 6 weeks training
  Number of participants that drop out from the study
Physical Activity Enjoyment Scale (PACES) score | Pre to post 6 weeks of home-based exergame training
  Change in Physical Activity Enjoyment Scale (PACES) score (an 18-item scale designed to measure physical activity enjoyment)
Situation Motivation Scale (SIMS) | Pre to post 6 weeks of home-based exergame training
  Change in Situation Motivation Scale (SIMS) score
Qualitative interviews | Following 6 weeks of training
  Overall experience determined through qualitative interviews
Immersive Experience Questionnaire (IEQ) | Following 6 weeks of training
  Immersive experience during home-based exergame sessions
Executive Functioning | Pre to post 6 weeks of home-based exergame training
  Change in reaction time determined using Test for Attentional Performance
Dynamic balance | Pre to post 6 weeks of home-based exergame training
  Change in dynamic balance determined using Y-Balance Test
Whole body adipose tissue | Pre to post 6 weeks of home-based exergame training
  Change in whole body adipose tissue volume using InBody body composition analyser
Visceral adipose tissue | Pre to post 6 weeks of home-based exergame training
  Change in visceral adipose tissue mass using InBody body composition analyser
Fat free mass | Pre to post 6 weeks of home-based exergame training
  Change in fat free mass using InBody body composition analyser
Blood pressure | Pre to post 6 weeks of home-based exergame training
  Change in blood pressure (systolic, diastolic and mean)
C-reactive protein | Pre to post 6 weeks of home-based exergame training
  Change in C-reactive protein
Total cholesterol | Pre to post 6 weeks of home-based exergame training
  Change in total cholesterol
Low Density Lipoprotein | Pre to post 6 weeks of home-based exergame training
  Change in low density lipoprotein
High Density Lipoprotein | Pre to post 6 weeks of home-based exergame training
  Change in high density lipoprotein
Triglycerides | Pre to post 6 weeks of home-based exergame training
  Change in triglycerides
HbA1c | Pre to post 6 weeks of home-based exergame training
  Change in HbA1c
Fasting glucose concentration | Pre to post 6 weeks of home-based exergame training
  Change in fasting glucose concentration
Fasting insulin concentration | Pre to post 6 weeks of home-based exergame training
  Change in fasting insulin concentration
Mean daily glucose concentration and area under the glucose curve | Pre to post 6 weeks of home-based exergame training
  Change in mean daily glucose concentration and area under the glucose curve
Coefficient of variation | Pre to post 6 weeks of home-based exergame training
  Change in coefficient of variation in continuous glucose monitor
Mean Daily steps | Pre to post 6 weeks of home-based exergame training
  Change in daily steps monitored by an accelerometer in percent

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amanat S, Ghahri S, Dianatinasab A, Fararouei M, Dianatinasab M. Exercise and Type 2 Diabetes. Adv Exp Med Biol. 2020;1228:91-105. doi: 10.1007/978-981-15-1792-1_6. PMID 32342452
- [Background] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Chtourou H, Trabelsi K, H'mida C, Boukhris O, Glenn JM, Brach M, Bentlage E, Bott N, Shephard RJ, Ammar A, Bragazzi NL. Staying Physically Active During the Quarantine and Self-Isolation Period for Controlling and Mitigating the COVID-19 Pandemic: A Systematic Overview of the Literature. Front Psychol. 2020 Aug 19;11:1708. doi: 10.3389/fpsyg.2020.01708. eCollection 2020. PMID 33013497
- [Background] Ding D, Lawson KD, Kolbe-Alexander TL, Finkelstein EA, Katzmarzyk PT, van Mechelen W, Pratt M; Lancet Physical Activity Series 2 Executive Committee. The economic burden of physical inactivity: a global analysis of major non-communicable diseases. Lancet. 2016 Sep 24;388(10051):1311-24. doi: 10.1016/S0140-6736(16)30383-X. Epub 2016 Jul 28. PMID 27475266
- [Background] Donath L, Roth R, Hurlimann C, Zahner L, Faude O. Pilates vs. Balance Training in Health Community-Dwelling Seniors: a 3-arm, Randomized Controlled Trial. Int J Sports Med. 2016 Mar;37(3):202-10. doi: 10.1055/s-0035-1559695. Epub 2015 Dec 2. PMID 26630547
- [Background] Franklin BA, Bonzheim K, Gordon S, Timmis GC. Safety of medically supervised outpatient cardiac rehabilitation exercise therapy: a 16-year follow-up. Chest. 1998 Sep;114(3):902-6. doi: 10.1378/chest.114.3.902. No abstract available. PMID 9743182
- [Background] Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL Jr, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC Jr; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). ACC/AHA 2002 guideline update for exercise testing: summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). Circulation. 2002 Oct 1;106(14):1883-92. doi: 10.1161/01.cir.0000034670.06526.15. No abstract available. PMID 12356646
- [Background] Gibbons RJ, Balady GJ, Beasley JW, Bricker JT, Duvernoy WF, Froelicher VF, Mark DB, Marwick TH, McCallister BD, Thompson PD Jr, Winters WL, Yanowitz FG, Ritchie JL, Gibbons RJ, Cheitlin MD, Eagle KA, Gardner TJ, Garson A Jr, Lewis RP, O'Rourke RA, Ryan TJ. ACC/AHA Guidelines for Exercise Testing. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Exercise Testing). J Am Coll Cardiol. 1997 Jul;30(1):260-311. doi: 10.1016/s0735-1097(97)00150-2. No abstract available. PMID 9207652
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Hallal PC, Andersen LB, Bull FC, Guthold R, Haskell W, Ekelund U; Lancet Physical Activity Series Working Group. Global physical activity levels: surveillance progress, pitfalls, and prospects. Lancet. 2012 Jul 21;380(9838):247-57. doi: 10.1016/S0140-6736(12)60646-1. PMID 22818937
- [Background] Jekauc D, Nigg C, Nigg CR, Reichert M, Krell-Roesch J, Oriwol D, Schmidt S, Wunsch K, Woll A. Measurement properties of the German version of the Physical Activity Enjoyment Scale for adults. PLoS One. 2020 Nov 18;15(11):e0242069. doi: 10.1371/journal.pone.0242069. eCollection 2020. PMID 33206685
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Morgan F, Battersby A, Weightman AL, Searchfield L, Turley R, Morgan H, Jagroo J, Ellis S. Adherence to exercise referral schemes by participants - what do providers and commissioners need to know? A systematic review of barriers and facilitators. BMC Public Health. 2016 Mar 5;16:227. doi: 10.1186/s12889-016-2882-7. PMID 26944952
- [Background] Motl RW, Dishman RK, Saunders R, Dowda M, Felton G, Pate RR. Measuring enjoyment of physical activity in adolescent girls. Am J Prev Med. 2001 Aug;21(2):110-7. doi: 10.1016/s0749-3797(01)00326-9. PMID 11457630
- [Background] Myers J. Cardiology patient pages. Exercise and cardiovascular health. Circulation. 2003 Jan 7;107(1):e2-5. doi: 10.1161/01.cir.0000048890.59383.8d. No abstract available. PMID 12515760
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Scott SN, Shepherd SO, Andrews RC, Narendran P, Purewal TS, Kinnafick F, Cuthbertson DJ, Atkinson-Goulding S, Noon T, Wagenmakers AJM, Cocks M. A Multidisciplinary Evaluation of a Virtually Supervised Home-Based High-Intensity Interval Training Intervention in People With Type 1 Diabetes. Diabetes Care. 2019 Dec;42(12):2330-2333. doi: 10.2337/dc19-0871. Epub 2019 Sep 17. PMID 31530660
- [Background] Scott SN, Shepherd SO, Hopkins N, Dawson EA, Strauss JA, Wright DJ, Cooper RG, Kumar P, Wagenmakers AJM, Cocks M. Home-hit improves muscle capillarisation and eNOS/NAD(P)Hoxidase protein ratio in obese individuals with elevated cardiovascular disease risk. J Physiol. 2019 Aug;597(16):4203-4225. doi: 10.1113/JP278062. Epub 2019 Jul 15. PMID 31218680
- [Background] Shepherd SO, Cocks M, Tipton KD, Ranasinghe AM, Barker TA, Burniston JG, Wagenmakers AJ, Shaw CS. Sprint interval and traditional endurance training increase net intramuscular triglyceride breakdown and expression of perilipin 2 and 5. J Physiol. 2013 Feb 1;591(3):657-75. doi: 10.1113/jphysiol.2012.240952. Epub 2012 Nov 5. PMID 23129790
- [Background] Tari AR, Nauman J, Zisko N, Skjellegrind HK, Bosnes I, Bergh S, Stensvold D, Selbaek G, Wisloff U. Temporal changes in cardiorespiratory fitness and risk of dementia incidence and mortality: a population-based prospective cohort study. Lancet Public Health. 2019 Nov;4(11):e565-e574. doi: 10.1016/S2468-2667(19)30183-5. PMID 31677775
- [Background] Trost SG, Owen N, Bauman AE, Sallis JF, Brown W. Correlates of adults' participation in physical activity: review and update. Med Sci Sports Exerc. 2002 Dec;34(12):1996-2001. doi: 10.1097/00005768-200212000-00020. PMID 12471307